CLINICAL TRIAL: NCT02697695
Title: Impact of Obesity and Metabolic Surgery on Chronic Inflammation
Brief Title: Chronic Inflammation After Obesity Surgery
Status: Completed | Type: Observational
Sponsor: Sana Klinikum Offenbach (Other)
Responsible Party: Principal Investigator, Sonja Chiappetta, MD, Dr. Sonja Chiappetta, Sana Klinikum Offenbach
Other Study IDs: FF 145/2015
Record Dates: First submitted 2016-02-20; First posted 2016-03-03 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Obesity
Keywords: chronic inflammation; fatty liver index
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- laparoscopic sleeve gastrectomy: patients who underwent laparoscopic sleeve gastrectomy (LSG) due to obesity and/or metabolic syndrome
  Interventions: Other: Laboratory Examination
- laparoscopic Roux-en-Y- gastric bypass: patients who underwent laparoscopic Roux-en-Y- gastric bypass (LRYGB) due to obesity and/or metabolic syndrome
  Interventions: Other: Laboratory Examination
- laparoscopic omega-loop gastric bypass: patients who underwent laparoscopic omega-loop gastric bypass (LOLGB) due to obesity and/or metabolic syndrome
  Interventions: Other: Laboratory Examination

INTERVENTIONS:
Other: Laboratory Examination — Laboratory Examination before, 1 month, 3 month, 6 month and up to 12 month after LSK, LRNYGB, LOLGB

SUMMARY:
To evaluate the impact of obesity surgery on chronic inflammation.

DETAILED DESCRIPTION:
A retrospective study to compare the impact of laparoscopic sleeve gastrectomy (LSG), laparoscopic Roux-en Y- gastric bypass (LRYGB) and laparoscopic omega-loop gastric bypass (LOLGB) on chronic inflammation and metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 35kg/m² and obesity-related disease or BMI > 40kg/m²

Exclusion Criteria:

* acute inflammation during laboratory examination

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent LSG, LRYGB, LOLGB due to obesity and/or metabolic syndrome
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Chronic inflammation | one day preoperatively, and 1 month, 3 month, 6 month and up to 12 month postoperatively
  the changing of leucocytes in /nl after obesity surgery

SECONDARY OUTCOMES:
Fatty liver index | one day preoperatively and 1 month, 3 month, 6 month and up to 12 month postoperatively
  the changing of fatty liver index after obesity surgery
Liver enzymes | one day preoperatively and 1 month, 3 month, 6 month and up to 12 month postoperatively
  the changing of GOT in U/l, GPT in U/l, GGT in U/l, AP in U/l after obesity surgery
Body Mass Index (BMI) in kg/m² | one day preoperatively and 1 month, 3 month, 6 month and up to 12 month postoperatively
  the changing of BMI in kg/m² before and after obesity surgery
weight in kg | one day preoperatively and 1 month, 3 month, 6 month and up to 12 month postoperatively
  the changing of weight before and after obesity surgery
waist circumference | one day preoperatively and 1 month, 3 month, 6 month and up to 12 month postoperatively
  the changing of waist circumference in cm before and after obesity surgery
HbA1c | one day preoperatively and 1 month, 3 month, 6 month and up to 12 month postoperatively
  the changing of HbA1c in % and after obesity surgery
Chronic inflammation II | one day preoperatively and 1 month, 3 month, 6 month and up to 12 month postoperatively
  the changing of c-reactive protein in mg/l after obesity surgery
Acute inflammation | one day preoperatively and one and four days postoperatively
  the changing of c-reactive protein in mg/l after obesity surgery
Acute inflammation II | one day preoperatively and one and four days postoperatively
  the changing of leucocytes in /nl after obesity surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Weiner, MD, Study Chair — Sana Klinikum Offenbach, Department of Obesity and Metabolic Surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hotamisligil GS. Inflammation and metabolic disorders. Nature. 2006 Dec 14;444(7121):860-7. doi: 10.1038/nature05485. PMID 17167474
- [Result] Nijhuis J, Rensen SS, Slaats Y, van Dielen FM, Buurman WA, Greve JW. Neutrophil activation in morbid obesity, chronic activation of acute inflammation. Obesity (Silver Spring). 2009 Nov;17(11):2014-8. doi: 10.1038/oby.2009.113. Epub 2009 Apr 23. PMID 19390527
- [Result] Morshed G, Fathy SM. Impact of post-laparoscopic sleeve gastrectomy weight loss on C-reactive protein, lipid profile and CA-125 in morbidly obese women. Wideochir Inne Tech Maloinwazyjne. 2016 Jan;10(4):521-6. doi: 10.5114/wiitm.2015.56480. Epub 2015 Dec 15. PMID 26865887
- [Result] Wellen KE, Hotamisligil GS. Inflammation, stress, and diabetes. J Clin Invest. 2005 May;115(5):1111-9. doi: 10.1172/JCI25102. PMID 15864338
- [Result] Furukawa S, Fujita T, Shimabukuro M, Iwaki M, Yamada Y, Nakajima Y, Nakayama O, Makishima M, Matsuda M, Shimomura I. Increased oxidative stress in obesity and its impact on metabolic syndrome. J Clin Invest. 2004 Dec;114(12):1752-61. doi: 10.1172/JCI21625. PMID 15599400
- [Derived] Chiappetta S, Schaack HM, Wolnerhannsen B, Stier C, Squillante S, Weiner RA. The Impact of Obesity and Metabolic Surgery on Chronic Inflammation. Obes Surg. 2018 Oct;28(10):3028-3040. doi: 10.1007/s11695-018-3320-y. PMID 29876839